CLINICAL TRIAL: NCT06394882
Title: FamCe-HLP- Family-centered Obesity Management Program in Primary Care Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Collaborators: Sultan Qaboos University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC/SR-CON/MCHH/22/02
Record Dates: First submitted 2023-12-06; First posted 2024-05-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity; Family; Behavior, Health; Lifestyle, Healthy
Keywords: childhood obesity; family; management; primary care
MeSH Terms: conditions — Pediatric Obesity; Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster Randomized controlled clinical trial to test the efficacy of a family-centered healthy lifestyle program on adiposity and weight status in mother-child dyads with overweight or obesity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The program will provide a seven-month program comprising two primary therapies: a three-month intensive behavioral therapy (IBT) and a four-month maintenance behavioral therapy (MBT). The three-month IBT will involve 12-week visits and exercise sessions. The program will encompass in-person (clinic/ health center) and online (telehealth) 12-weekly visits. The 60-minute consultations and booster sessions will be provided by a qualified multidisciplinary team (obesity nurse, psychologist, nutritionist, and physiotherapist), each consulting in their expertise. In collaboration with the physical education and sports science department at Sultan Qaboos University, mothers in the intervention group will be provided exercise sessions based on their individual metabolic and physiological parameters. The maintenance behavioral therapy will start one month after the end of the IBT and will involve four monthly support meetings on a group level.
  Interventions: Behavioral: Family-Centered Healthy Lifestyle Program (FamCe-HLP)
- Treatment as usual (No Intervention): Participants in the control group will receive treatment as usual, which is the regular care provided by the center for adults and children with obesity.

INTERVENTIONS:
Behavioral: Family-Centered Healthy Lifestyle Program (FamCe-HLP) — A multidisciplinary-led healthy lifestyle program will provide a seven-month program comprising two primary therapies: a three-month intensive behavioral therapy (IBT) and a four-month maintenance behavioral therapy (MBT). The program will run on scheduled days using one of the center's offices for the IBT and the center's seminar room for the MBT.
  Arms: Intervention Group

SUMMARY:
This clinical trial aims to compare the adiposity and weight status among mother-child dyads with overweight or obesity who receive the Fam-Ce-HLP intervention with the mother-child dyads with overweight or obesity who did not receive the intervention. The main question[s] it aims to answer are:

* Is there a significant difference in the adiposity and weight status of mother-child dyads with overweight or obesity who received the Fam-Ce-HLP intervention compared with the mother-child dyads with overweight or obesity who did not receive the intervention?
* Is there a significant difference in the health behaviors, obesity stage level, and ripple effect of mother-child dyads with overweight or obesity who received the Fam-Ce-HLP intervention compared with the mother-child dyads with overweight or obesity who did not receive the intervention? Participants will be asked to attend a seven-month program comprising two primary therapies: a three-month intensive behavioral therapy (IBT) and a four-month maintenance behavioral therapy (MBT).

Researchers will compare the intervention group with the treatment-as-usual group (control group) to see if there is a difference in adiposity, weight status, health behaviors, obesity stage level, and ripple effect.

ELIGIBILITY:
Inclusion Criteria:

* Mother and child dyads with the presence of overweight or obesity (stages 0 to 2)
* Being Omani
* Mother age 18 years or more
* Child age 6 to 12 years
* Mother understand, write, and read in Arabic
* Eligible to receive the health center's services based on their area of residence
* Has medical clearance to participate in individual exercise sessions
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Mother or child currently receiving an obesity-related program
* Mother or child currently on obesity-related procedures
* Mother or child with a history of obesity-related surgeries in the last 5 years
* Mother or child is in obesity stage 3 or 4 based on the Edmonton obesity staging system
* Mother who is pregnant during the study time

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-06-21 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Child's Adiposity | Four time points in one year duration
  Child's body fat percentage will be determined through a bioelectrical impedance analysis scale
Mother's Adiposity (Body fat percentage) | Four time points in one year duration
  Mother's body fat percentage will be determined through a bioelectrical impedance analysis scale
Child's weight status (BMI z score) | Four time points in one year duration
  Child's weight and height will be combined to report BMI in kg/m^2 and then BMI z-scores will be determined according to the 2007 World Health Organization growth charts
Mother's weight status (BMI) | Four time points in one year duration
  Mother's weight and height will be combined to report BMI in kg/m^2

SECONDARY OUTCOMES:
Child's daily caloric intake in kilocalories (24 dietary recall) | Four time points in one year duration
  Child's 24 dietary recall for three non-consecutive days will be collected using myfood24 nutritional analysis software
Child's food frequency intake of main food groups in grams (grains, fruits, vegetables, dairy, protein) | Two time points in one year
  Child's food frequency of main food groups will be assessed through a semiquantitative food frequency questionnaire (FFQ)
Mother's food frequency intake of main food groups in grams (grains, fruits, vegetables, dairy, protein) | Two time points in one year
  Mother's food frequency of main food groups will be assessed through a semiquantitative food frequency questionnaire (FFQ)
Child's moderate to vigorous physical activity in minutes per day | Four time points in one year duration
  Child's physical activity level will be determined through calculating the moderate to vigorous physical activity in minutes per day by wearing accelerometers (Actigraph devices) for seven days
Mother's moderate to vigorous physical activity in minutes per day | Four time points in one year duration
  Mother's physical activity level will be determined through calculating the moderate to vigorous physical activity in minutes per day by wearing accelerometers (Actigraph devices) for seven days
Child's obesity stage level | Four time points in one year duration
  Child's obesity stage level will be assessed following the Edmonton obesity staging system evaluation by a family physician
Mother's obesity stage level | Four time points in one year duration
  Mother's obesity stage level will be assessed following the Edmonton obesity staging system evaluation by a family physician
Father's weight status (ripple effect | Four time points in one year duration
  Father's weight and height will be combined to report BMI in kg/m^2
Child's 18 and above years old sibling weight status (ripple effect) | Four time points in one year duration
  Child's over 18 years old sibling weight and height will be combined to report BMI in kg/m^2
Child's under 18 years old sibling weight status (ripple effect) | Four time points in one year duration
  Child's under 18 years old sibling weight and height will be combined to report BMI in kg/m^2 and then BMI z-scores will be determined according to the 2007 World Health Organization growth charts

CONTACTS AND LOCATIONS:
Overall Officials: Basma Al Yazeedi, PhD, Principal Investigator — Sultan Qaboos University
Locations (4):
- Oman (4):
  - Mabela Health Center, Muscat, Muḩāfaz̧at Masqaţ
  - Mabela South Health Center, Muscat, Muḩāfaz̧at Masqaţ
  - Mawaleh Health Center, Muscat, Muḩāfaz̧at Masqaţ
  - Mawaleh North Health Center, Muscat, Muḩāfaz̧at Masqaţ

IPD SHARING:
Plan to Share IPD: No